CLINICAL TRIAL: NCT05545228
Title: A Randomised Feasibility Trial of an Intervention Using Mental Health Support Workers as Link Workers to Improve Dental Visiting in People With Severe Mental Illness: The Mouth in Mind Study
Brief Title: The Mouth Matters in Mental Health Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Jasper Palmier-Claus, Principle Investigator, Lancaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRAS304696; NIHR132853 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2022-09-08; First posted 2022-09-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Mental Disorders, Severe
Keywords: Mental Health; Oral Health; Dentistry
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A feasibility single-blinded randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive treatment as usual plus a link work intervention to support access to dental services.
  Interventions: Behavioral: Link work intervention
- Treatment as usual group (No Intervention): Participants to receive treatment as usual and will not receive the intervention.

INTERVENTIONS:
Behavioral: Link work intervention — Intervention from a link worker to support participants to access dental services.
  Arms: Intervention group

SUMMARY:
To investigate the feasibility and acceptability of a link work intervention to increase planned dental care visits for patients with severe mental illness, and through this to improve their oral health.

1. To understand what constitutes best practice when delivering link work around dental visiting.
2. To identify what training needs exist for support workers around link work.
3. To determine whether patients with SMI are willing to be randomised to a trial targeting dental visiting.
4. To understand whether it is feasible to collect clinical outcome and planned dental appointment data in this population.
5. To explore if, and how, patients with severe mental illness engage with a link work intervention.
6. To understand the potential factors impacting (e.g. facilitators and barriers) acceptability and delivery.

DETAILED DESCRIPTION:
Background and study aims

Severe mental ill health (SMI) affects around 1% of the population. It includes depression, psychosis, and bipolar disorder. People with experience of SMI are more likely to have problems with their teeth and gums. This includes more missing, filled, and decayed teeth than people without SMI. Having poor oral health can impact a lot of everyday activities like eating, speaking and smiling. It can affect how patients see themselves and their mental health.

Dentists can treat many early teeth and gum problems. However, very few people with SMI attend regular dental appointments. Instead, they are more likely to seek help when in crisis and invasive treatments are the only option. Accessing a dentist for people with SMI can be difficult for lots of reasons. People can feel helpless, fearful, or unmotivated to attend. They can have difficulty booking, planning, and getting to appointments. They may struggle to pay for or access free dental care. Unfortunately, existing dental initiatives have not addressed the barriers facing this group. They do not help people with SMI to attend the dentist.

The investigators want to help people with SMI to access dental care. The study will use mental health support workers who are already working in the National Health Service (NHS). They will link people receiving care from mental health teams with dental services. The support workers will help people to book, plan, and attend regular dental appointments. They will support patients to apply for financial support. People call this type of support link work. Research has indicated that link work can increase dental visits in people who might not normally attend. Mental health support workers already do link work for other appointments. Link work has been used to help other vulnerable groups of people (e.g. children) around dental care. However, this will be the first use of link work to help people with SMI to attend the dentist.

Who can participate?

People with a severe mental health difficulties currently accessing secondary care mental health services at the point of referral (e.g. community mental health team, early intervention for psychosis service), but who have not had a routine dental appointment in the past three years.

What does the study involve?

Participants will be randomly allocated to receiving treatment as usual or treatment as usual plus the link work intervention. This will be decided by chance. The investigators will measure how often people in both groups visit the dentist. They will also assess the state of their teeth and gums. They will collect this data when people come into the study and after nine months. The authors will offer interviews to patients and staff involved in the trial to understand how they found their involvement.

What are the possible benefits and risks of participating?

The intervention aims to support people to access dental services. However, it is currently untested, which is the reason for doing the research.

When is the study starting and how long it is expected to run for?

Recruitment for the trial is starting in September 2022 and will run for seven months. The whole project is scheduled to finish in April 2024.

Who is funding the study?

The National Institute of Health Research (NIHR) Health and Social Care Delivery Research (HS&DR) scheme are funding the project.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >18 years
2. Able to provide informed consent
3. Receipt of care from a Community Mental Health Team (or equivalent service) or Early Intervention Team at the point of referral
4. No routine and planned dental appointment in the past 3 years. The person should not have accessed a dental service (e.g. high street dentist, special care dentist service) for routine or planned dental care in the past 3 years. This would include any dental examination, diagnosis, advice or treatment (e.g. fillings, root canal, extractions, crowns, dentures, bridges) resulting from a routine (non-emergency) appointment at a dental service. The researchers do not consider emergency dental care (e.g. attendance at A&E, dental hospital) within this definition, although any follow-up routine and planned appointments with a dentist would exclude the person from taking part.

Exclusion criteria:

1. Inpatient status on a psychiatric or secure ward. The researchers will allow participants in supported living to take part as long as they are in receipt of care from a Community Mental Health Team (or equivalent service) or Early Intervention for Psychosis Service
2. Immediate risk to self or others operationalised as the presence of active intent or planning to harm oneself or others in the near future (e.g. next month). Where individuals are excluded on this basis, with the person's consent, the researcher will aim to re-contact them and the referrer in approximately 1 month's time (or a time period agreed in collaboration with the individual) to determine if the risk has subsided to a point where they are now eligible.
3. Enrolled in a dental trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates - feasibility criteria | 7 months
  Data on ability to recruit randomise 84 participants to target in a 7-month recruitment window. Green ≥80%. Amber 60-79%. Red ≤59%.
Visiting data - feasibility criteria | 9 months
  Percentage of participants with available data on dental visiting via self-report or BSA data. Green ≥90%. Amber 60-89%. Red ≤59%.
Clinical exam - feasibility criteria | 9 months
  Percentage of participants completing the dental examination. Green ≥80%. Amber 60-79%. Red: ≤59%.
Adherence to intervention - feasibility criteria | 9 months
  Percentage of participants receiving intervention ≥1 sessions during nine month window. Green ≥80%. Amber 60-79%. Red ≤59%.
Intervention and trial protocol - feasibility criteria | 9 months
  Qualitative data to understand the acceptability and feasibility of the procedures, assessments, and intervention to inform a full trial and service delivery. This will be via qualitative interviews with service users (participants), research staff (link workers, research assistants), and key stakeholders (referrers, managers, commissioners). Audio recordings of sessions and field notes will also be analysed.
Safety of intervention - feasibility criteria | 9 Months
  Monitoring and review of research related serious adverse events (SAEs). The Trial Steering Committee (TSC) will oversee SAEs across treatment arms. The authors will discontinue the trial if the intervention or procedures elevate risk.

SECONDARY OUTCOMES:
Brief Pain Inventory - short form | Baseline and 9 month assessments
  A questionnaire to assess orofacial pain.
Manchester Orofacial Pain Disability Scale | Baseline and 9 month assessments
  Pain related disability
Oral Health Impact Profile | Baseline and 9 month assessments
  Oral health related quality of life
Confidence around dental visiting | Baseline and 9 month assessments
  Item asking about confidence in visiting the dentist. "How confident are you that you will be able to attend a dental appointment?" (1, no confident; 7, very confident)
Rosenberg Self-esteem Scale (RSES) | Baseline and 9 month assessments
  Assessing self-esteem
Modified Dental Anxiety Scale | Baseline and 9 month assessments
  Assessing dental anxiety
Patient Health Questionnaire (PHQ) | Baseline and 9 month assessments
  Assessing depression
EuroQol 5 Dimension (EQ-5D-5L) | Baseline and 9 month assessments
  Assessing quality of life
The number of eligible participants able to access free or subsidised dental care | Baseline and 9 month assessments
  Assessing ability to successfully access free or subsidised dental care collected via the business services authority and self-report.
The number of planned dental appointments attended | Baseline and 9 month assessments
  The research team will record and report the number of routine dental appointments attended, recorded by both the business services authority and self-report.
Oral health self-management - tooth brushing, mouth wash, and flossing | Baseline and 9 month assessments
  'How often do you brush your teeth nowadays?' (ordinal five-point scale); 'How long do you brush your teeth for nowadays?' (ordinal five-point scale); 'How often do you clean between your teeth (inter-dental cleaning with floss, inter-dental brushes, tooth picks)?' (ordinal five-point scale); and 'Do you use a fluoride mouth-wash?' (binary)
Self reported attendance at a planned dental appointment | 9 months
  The research team will ask people the following 'Have you attended a dental service since the baseline assessment (nine months ago)? This would include a routine appointment with a dentist or special care dentistry service. It could also include a planned appointment at a dental hospital. However, it would not include an emergency dental appointment.'. Participants will also be asked to provide the dates and times of dental appointments. This outcome will be coded as whether the person has or has not accessed a planned dental appointment via self-report.
Business services authority recorded attendance at a planned dental appointment | 9 months
  NHS England collects information on visiting behaviour via the Business Services Authority. The research team will gain participants consent to extract this data, which the researchers will then match to the participants research data. The business services authority will be used to collect data on whether a planned care appointment has taken place. This data will only pick up National Health Service, and not private, dental appointments. This outcome will be coded as whether the person has or has not accessed a planned dental appointment via the business services authority data.
Number of decayed, missing, or filled teeth (DMFT) via dental examination | Baseline and 9 months
  An examination for dental caries in permanent teeth will involve examining 32 teeth (i.e. all permanent teeth including wisdom teeth) with a metallic periodontal probe (Community Periodontal Index (CPI) probe) and a plane mouth mirror.
Pulpal involvement, ulceration due to trauma, fistula, and abscess (PUFA) via dental examination | Baseline and 9 months
  The PUFA score per person is calculated in the same cumulative way as for the DMFT and represents the number of teeth that meet the PUFA diagnostic criteria. Thus, for an adult in our study the score can range from 0 to 32 PUFA.
Modified Plaque Score via dental examination | Baseline and 9 months
  The locally derived system involves assessing six teeth representative of the entire dentition, for the worst plaque score on each tooth surface from visual examination and, where necessary, the use of a probe to detect the presence of plaque. These six teeth are the UL4 UL1 UR6 LL6 LR1 LR4. Each surface; Interproximal, buccal and lingual or palatal of the six teeth should be viewed in turn and the highest level of visible plaque on each surface should be scored '2'.

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Palmier-Claus, PhD, DClinPsy, Principal Investigator — Lancaster University; Rebecca Harris, BDS, PhD, Principal Investigator — University of Liverpool
Locations (5):
- United Kingdom (5):
  - Pennine Care NHS Foundation Trust, Ashton-under-Lyne, Great Manchester
  - Greater Manchester Mental Health NHS Foundation Trust, Manchester, Great Manchester
  - University of Manchester, Manchester, Greater Manchester
  - Lancaster University, Lancaster, Lancashire
  - Lancashire and South Cumbria NHS Foundation Trust, Preston, Lancashire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmier-Claus J, Morris A, French P, Griffiths R, Aggarwal VR, Berry K, Gkioni E, Harris R, Laverty L, Lobban F, Procter S, Kerry E, Newens C, Mupinga P, Golby R, Valemis K, Oakes L, Fazekas F, Perry A, Shiers D, Lodge C, Hilton C, Dawber A, Elliott E, Lunat F, Burnside G. A Link Work Intervention to Facilitate Dental Visiting in People With Severe Mental Illness: A Two-Arm, Multi-Site, Assessor Blind, Randomised Feasibility Trial With Dental Record Linkage. Community Dent Oral Epidemiol. 2025 Oct;53(5):580-586. doi: 10.1111/cdoe.70002. Epub 2025 Aug 4. PMID 40755121
- [Derived] Hilton C, Morris A, Burnside G, Harris R, Aggarwal VR, Procter S, Griffiths R, French P, Laverty L, Lobban F, Berry K, Shiers D, Golby R, Fazekas F, Valemis K, Perry A, Newens C, Kerry E, Mupinga P, Gkioni E, Lodge C, Dawber A, Elliott E, Lunat F, Palmier-Claus J. A two-arm, randomised feasibility trial using link workers to improve dental visiting in people with severe mental illness: a protocol paper. Pilot Feasibility Stud. 2023 Sep 8;9(1):157. doi: 10.1186/s40814-023-01383-2. PMID 37684682
- See also: Trial website — https://www.lancaster.ac.uk/health-and-medicine/research/spectrum/research/the-mouth-matters-in-mental-health-study/

DOCUMENTS (2):
  • Study Protocol (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT05545228/Prot_001.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT05545228/SAP_002.pdf